CLINICAL TRIAL: NCT02435498
Title: A Web-based Education Module Versus Standard of Care for Pain Management Following a Fracture in Children: a Randomized Controlled Trial
Brief Title: Web-based Education Module for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Naveen Poonai, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 106402
Record Dates: First submitted 2015-04-29; First posted 2015-05-06 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Bone Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Videotape Recording; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Interactive website (Experimental): The interactive website called Online User Centered Home Pain Management for Fractures (OUCH PMF) will cover 4 domains of knowledge: 1. Fracture-related pain 2. Analgesic dosing regimens 3. Indications, risks and safety of analgesia in children 4. Signs and symptoms of pain in children
  Interventions: Other: Interactive website
- Video (Active Comparator): The online video will contain the same information within the website.
  Interventions: Other: Video
- Standard of care (Active Comparator): Standard of care includes a pamphlet with cast care instructions and verbal instructions on caring for the child at home.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Interactive website — The interactive website called Online User Centered Home Pain Management for Fractures (OUCH PMF) will cover 4 domains of knowledge: 1. Fracture-related pain 2. Analgesic dosing regimens 3. Indications, risks and safety of analgesia in children 4. Signs and symptoms of pain in children
  Arms: Interactive website
Other: Video — The online video will contain the same information within the website.
  Arms: Video
Other: Standard of care — Standard of care includes a pamphlet with cast care instructions and verbal instructions on caring for the child at home.
  Arms: Standard of care

SUMMARY:
This study's objectives are as follows:

1. To evaluate the utility of a website to provide information and guidance about pain management in children 2. To educate parents about the pathophysiology of pain, proper use of analgesic medications and signs of pain in children 3. To reduce the functional impact of pain in children following treatment for fracture 4. To endow parents with confidence to manage their child's pain at home 5. To dispel misconceptions about the use and safety of analgesics in children 6. To increase awareness of complications of fractures such as compartment syndrome

DETAILED DESCRIPTION:
This study will compare the effectiveness of three mediums of parental education among parents of children treated for non-operative fractures in the emergency department (ED): 1) A novel website entitled, "Online User-Centered Home Pain Management for Fractures" (OUCH PMF) 2) An online educational video (OV) and 3) standard discharge instructions (SOC). The investigators primary goal is to see which modality results in a greater improvement in scores on a on a knowledge questionnaire. The investigators secondary goals are to see which modality results in better parental satisfaction, confidence in managing pain, and lower impact of injury on the child and family. As participants will receive the standard-of-care that includes a pamphlet on how to take care of the cast. During their stay in the ED, participants will be randomly assigned to one of the three aforementioned groups. Participants will then be given the pre-intervention knowledge questionnaire, followed by the intervention and then the post-intervention knowledge questionnaire, prior to being discharged. At 120 hours post-discharge, participants will be asked to access an online survey to obtain information about the functional impact of the injury on their child. The investigators goal is to compare online and video education tools in their ability to improve parental knowledge, confidence, and satisfaction regarding the treatment of fracture pain.

ELIGIBILITY:
Inclusion Criteria:

* All caregivers who are in attendance with their child (any age) for a primary complaint of a non-operative fracture managed by the paediatric emergency physician AND will be the primary caregiver for the child at home.

Exclusion Criteria:

* Poor parental English fluency
* Lack of a home computer with Internet access
* Child with a history of renal disease, liver disease, bleeding diathesis, chronic pain issues, or pregnancy.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change in 21-item knowledge questionnaire total score between groups | 120 hours

SECONDARY OUTCOMES:
Number of days of work missed for parent | 120 hours
Parental confidence in recognizing pain and providing analgesia using a 5-point Likert scale | 120 hours
Number of sleep-interrupted nights for child | 120 hours
Number of days of school missed for child | 120 hours
Number of days before resumption of normal diet for child | 120 hours
Other educational resources used | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, Principal Investigator — Western University
Locations (1):
- Children's Hospital, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No